CLINICAL TRIAL: NCT00586677
Title: Evaluation of Parenting Interventions to Decrease Family Risk for Child
Brief Title: Evaluation of Parenting Interventions to Decrease Family Risk for Child Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00016431; 7194 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Child Abuse
Keywords: child abuse; child neglect; PCIT; Lutzker; attachment; parenting
MeSH Terms: interventions — Health; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RF (Active Comparator): Relationship focused where the primary goals are to strengthen the relationship between the parent and the child and to give the parent additional skills that can be used to manage the behavior of the child.
  Interventions: Behavioral: Parent-Child Interaction Therapy; Behavioral: Early Relationships
- HS (Active Comparator): The physical health and safety are the primary components of this parenting program where the parent is taught about basic healthcare and safety in the home.
  Interventions: Behavioral: Health and Safety

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy — Sixteen one hour sessions done in-home for children ages 2-7. Proceed through protocol based on mastery of predefined skills.
  Other Names: PCIT
  Arms: RF
Behavioral: Health and Safety — Sixteen one hour sessions for children age 0-7 conducted in the home. Participants are quizzed on material to determine mastery.
  Arms: HS
Behavioral: Early Relationships — Sixteen one-hour sessions for children age 0-2 provided in-home.
  Arms: RF

SUMMARY:
The purpose of this research is to evaluate specific parenting programs that aim to improve the family's ability to keep children physically safe and emotionally secure. We would like to learn more about how the treatments actually help families and to find out how an intervention that focuses on child health and safety compares with one that focuses on the parent and child relationship. We also want to determine whether participating in one program type versus the other results in further reports for child maltreatment.

ELIGIBILITY:
Inclusion Criteria:

* resident of Durham, NC
* a child between the ages of 0-7 was the focus of the Department of Social Services report
* child's caregiver was the focus of the report
* Child Protective Services report occurred on or after June 1, 2004
* family is English speaking
* Sexual abuse was not "confirmed" or "highly suspicious" during an evaluation

Exclusion Criteria:

* Child Protective Services report of sexual abuse that was "confirmed" or "highly suspicious"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2005-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Durham County, North Carolina Department of Social Services accepted reports of child maltreatment | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dodge, Ph.D., Principal Investigator — Duke University; Karen O'Donnell, Ph.D., Principal Investigator — Duke University
Locations (1):
- Center for Child and Family Health, Durham, North Carolina, United States